CLINICAL TRIAL: NCT00850616
Title: A Phase I Dose Ranging Study of the Safety, Tolerability, and Immunogenicity of a 3-Dose Regimen of the MRKAd5 HIV-1 Trigene and the MRKAd6 HIV-1 Trigene Vaccines Alone and in Combination in Healthy Adults
Brief Title: Three-Dose Regimen of MRKAd5+6 Trigene (V526) in Healthy Adults (V526-001)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V526-001; 2009_551
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: HIV; HIV Infections
Keywords: HIV; HIV Seronegativity; Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- 1 (Experimental): MRKAd6 Trigene 0.5x10^9 Ad6 vg
  Interventions: Biological: V526
- 2 (Experimental): MRKAd6 Trigene 0.5x10^10 Ad6 vg
  Interventions: Biological: V526
- 3 (Experimental): MRKAd6 Trigene 0.5x10^11 Ad6 vg
  Interventions: Biological: V526
- 4 (Experimental): MRKAd5 Trigene 0.5x10^10 Ad5 vg
  Interventions: Biological: V526
- 5 (Experimental): MRKAd5 Trivalent 1.5x10^10 Ad5 vg
  Interventions: Biological: V526
- 6 (Experimental): MRKAd5+6 Trigene 1x10^9 Ad vg
  Interventions: Biological: V526
- 7 (Experimental): MRKAd5+6 Trigene 1x10^10 Ad vg
  Interventions: Biological: V526
- 8 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo to V526

INTERVENTIONS:
Biological: V526 — 0.5 mL intramuscular injections of MRKAd5+6 trigene vaccine (V526) in a 3-dose regimen on Day 1, Week 4 and Week 26.
  Arms: 1; 2; 3; 4; 5; 6; 7
Biological: Comparator: Placebo to V526 — 0.5 mL intramuscular injections of placebo to MRKAd5+6 trigene vaccine (V526) in a 3-dose regimen on Day 1, Week 4, and Week 26.
  Arms: 8

SUMMARY:
A study to assess the general safety and tolerability of the administration of the 3-dose regimen of the MRKAd5+6 trigene vaccine

ELIGIBILITY:
Inclusion Criteria:

* Subject has negative tests for HIV, Hepatitis B, and Hepatitis C within 60 days of injection
* Subject agrees to use an acceptable method of birth control through week 52 of the study

Exclusion Criteria:

* Subject has been given immune globulin or blood products within 30 days of first dose of study vaccine
* Subject has been vaccinated with a live virus vaccine within 30 days or an inactivated vaccine within 5 days of first dose of study vaccine
* Subject has known or suspected impaired immune function
* Subject has participated in any other HIV vaccine trial
* Female subject is pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2005-04; Primary Completion 2006-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 3-dose regimen of MRKAd5+6 trigene vaccine as assessed by review of AEs | Week 30
Immune response to MRKAd5+6 trigene vaccine | 30 week

SECONDARY OUTCOMES:
Immune response to MRKAd5+6 trigene vaccine in subjects with preexisting antibodies to Ad5 or Ad6 | Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Harro C, Sun X, Stek JE, Leavitt RY, Mehrotra DV, Wang F, Bett AJ, Casimiro DR, Shiver JW, DiNubile MJ, Quirk E; Merck V526-001 Study Group. Safety and immunogenicity of the Merck adenovirus serotype 5 (MRKAd5) and MRKAd6 human immunodeficiency virus type 1 trigene vaccines alone and in combination in healthy adults. Clin Vaccine Immunol. 2009 Sep;16(9):1285-92. doi: 10.1128/CVI.00144-09. Epub 2009 Jul 15. PMID 19605598